CLINICAL TRIAL: NCT02760537
Title: Lay Health Worker Model to Reduce Liver Cancer Disparities in Asian Americans
Acronym: LHWAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HopkinsIRB-00004537; 5R01CA163805-02 (NIH); JT 7061 (Other: JeffTrial Number)
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Liver Neoplasms; Hepatitis B
Keywords: Liver Neoplasms; Hepatitis B; Hepatitis B vaccination; Asian Americans; Lay health workers; Community health workers
MeSH Terms: conditions — Liver Neoplasms; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lay Health Worker Intervention (Experimental): LHWs conducted phone interventions by reminding participants of a series of vaccinations at months 1, 2, and 5 among those assigned to the intervention group. Those who had health insurance were encouraged to complete vaccinations through their providers. If participants did not have health insurance, LHWs provided resources to help those in the intervention access vaccinations by referring them to free vaccine events in the community.
  Interventions: Behavioral: Lay Health Worker Intervention
- Placebo (a list of resources) (Placebo Comparator): Those in the control group received a list of resources along with their results by mail that offered free vaccinations, such as local health departments.
  Interventions: Behavioral: Placebo (a list of resources)

INTERVENTIONS:
Behavioral: Lay Health Worker Intervention — Lay Health Worker Phone Intervention The second phase addressed phone intervention training, where LHWs who had completed the first phase and were willing to participate in the second phase learned the process for calling participants to remind them to complete a series of HBV vaccinations. The LHWs assigned to the intervention group conducted phone interventions by reminding participants about completing a series of vaccinations at Months 1, 2, and 6, and also provided accompanying resources and support.
  Arms: Lay Health Worker Intervention
Behavioral: Placebo (a list of resources) — Those in the control group received a list of resources along with their results by mail that offered free vaccinations, such as local health departments.
  Arms: Placebo (a list of resources)

SUMMARY:
The study was conducted between April 2013 and October 2014. In the parent study, 600 foreign-born Asian American adults 18 years of age and older were drawn from the community in the Baltimore Washington Metropolitan Area. Using a non-probability sampling method, foreign-born Asian American adults, 18 years of age and older, were recruited from the community.

After providing informed consent, all the participants were asked to complete a self-administered questionnaire in English, Chinese, Korean, or Vietnamese with the assistance of a bilingual interviewer when necessary. Then, all of the participants were instructed and given 5 to 10 to minutes to read culturally integrated and linguistically appropriate educational material (e.g., Photo novel) developed and validated for efficacy from a prior study.

All participants received hepatitis B testing: HBsAg (hepatitis B surface antigen), HBsAb (hepatitis B surface antibody) and, HBcAb (hepatitis B core antibody). A total of 600 completed the survey and screening. A week later, they received the results of the screening test. Based on the screening results, all participants were categorized into three groups: (1) infected (HbsAg+), (2) unprotected (HbsAg-/HbsAb-), or (3) protected (HbsAg-/HbsAb+). We sent the results by mail to participants who were unprotected and protected. Among those 600 screened participants, 33(5.5%) had chronic hepatitis B virus (HBV) infection and 335 (55.8%) had evidence of resolved HBV infection (protected). A total of 232 (38.7%) were susceptible to HBV infection (unprotected).

LHW (lay health worker) Intervention for those unprotected: Those unprotected (n=232) were randomly assigned to either the intervention (n=124) or the control (n=108) groups by computer-automated random assignment. Randomization was used to assure equivalence between groups on key factors that may potentially influence the outcome of HBV vaccinations: gender, age, education, length of stay in the U.S.

LHWs conducted phone interventions by reminding participants of a series of vaccinations at months 1, 2, and 5 among those assigned to the intervention group. Those in the control group received a list of resources along with their results by mail that offered free vaccinations, such as local health departments. Seven months after mailing the results, those unprotected were followed up by phone to ask about their status of the series of vaccinations and about promoters or barriers to vaccinations.

DETAILED DESCRIPTION:
Specific Aim 1. Develop a training protocol and certification program for lay health workers (LHWs)

People of Asian backgrounds are likely to exhibit cultural relativism leaning toward collectivism compared to individualism. The personal interactions within their self-identified cultural communities may closely relate to development of their perceived beliefs and subjective norms, which influence to act upon identified health behaviors (Ajzen, Albarracin & Hornik 2007). The investigators will develop a lay health worker (LHW) model that highlights the effects of culturally competent human and educational interactions on facilitating the Chinese-, Korean- and Vietnamese-American (CKV-A) community's active behaviors in hepatitis B screening, vaccination, and treatments. To develop an efficacious and effective LHW intervention that will contribute for creating a critical mass toward sustainable Chinese, Korean and Vietnamese (CKV) changes, our strategic approaches include as follows:

1. Review the liver cancer education program guidebook in English, (developed by previous project R25).
2. Refine/revise the approaches through work group reviews: Through a series of bi-monthly meetings with participants from community advisory board (CAB), CKV-A communities, health practitioners and outreach workers, and experts in hepatitis B virus (HBV) and liver cancer education (Juon and Lee), and education and evaluation (Park), the investigators will confirm/specify the approaches of the available materials and develop additional assessment approaches and forms in English.
3. Test the validities of subgroup language versions with pilot CKV groups: Through assessments with each group (n=10) of CKV-As, the investigators will produce the refined validated LHW protocol (after translation and back-translation). It will include common and unique approaches across/within subgroup(s) to be congruent with cultural values.
4. Test the pilot LHW implementation
5. Establish the LHW model to certify satisfactory practicum experience in Patient Navigation training module: Through ongoing assessments with the study participants and participating health care systems, the investigators will monitor the LHW experiential learning module to provide patient navigation function. The approach will identify barriers to hinder access to timely screening, follow-up, and treatment upon diagnosis.

Recruitment: Earp et al. (1997) suggest effective LHWs would have some or all of the following characteristics and skills: (1) the ability to comfortably and effectively access the health care system; (2) the ability to balance the demands of lay helping with other life responsibilities; (3) an interest in AA's health and social issues; (4) maintain close, supportive, and reciprocal connections with others; and (5) leadership skills. LHW models depend on genuine natural helpers to function. To increase recruitment potential for CKVs having desired characteristics: First, the investigators will reach a broad pool of adult volunteers, regardless of gender, income level, or health care experience, who have these characteristics and also have the ability to speak, read and write Chinese, Korean, or Vietnamese languages at or above 2nd grade level. Second, adopting a referral recruitment strategy in social market theory (Lefebvre et al. 1988) as it may be more effective for people who may be more responsive to their sense of collective cultural group's interactions, the investigators will recruit the first 10 LHW candidates per each ethnic group referred by word of mouth, faith-based organization leaders, community advisory groups, and health and social service agencies. Finally, the investigators will expand our recruitment continuously in the community. In Year 1, the investigators plan to train a total of 60 certified LHWs (20 from each ethnic group). The investigators estimate retention of 40 (67%) certified LHWs at the end of the Year 1, based upon literature reviews (Anderson 2000; Caulfield et al. 1998; Han et al. 2009). To replace drop-out LHWs in subsequent years, the investigators plan to recruit and train a total of 30 additional LHWs (10 for each ethnic group) from Years 2 to 3.

Process Evaluation: Using evaluation model of Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) (Glasgow et al. 2001), a framework that emphasized on Reach, Effectiveness, Adoption, Implementation and Maintenance, the investigators will examine the extent to which the LHW program is carried out through processes as intended. At individual level, the investigators will focus on Reach (R) of the LHW certification program and hepatitis B free events and on the Efficacy/Effectiveness (E) of the LHW certification program. For the group level of aggregated individuals, the investigators will assess on Adoption (A), Implementation (I), and Maintenance (M). The investigators will assess general administrative processes of LHW program during the study period in the selected perspectives of fidelity (e.g. logistic reviews, completion rates), dose (e.g. satisfaction survey), and method on translated forms and tools (Saunders, Evans, & Joshi 2005).

Specific Aim 2. To assess the prevalence of HBV infection by providing screening test

A total of 600 Asian American adults (200 Chinese, Koreans, and Vietnamese each), 18 years of age and older will be drawn from the community.

Recruitment strategy. The investigators have two major channels to recruit participants with the help of certified LHWs including hepatitis B initiative of Washington DC (HBI-DC) screening events and Asian American Health Center (AAHC). First, in the past 10 years, the HBI-DC has screened over 3000 individuals in the Baltimore-Washington Metropolitan Area and approximately 8 to 11% are positive for the surface antigen of the hepatitis B virus (HBsAg). Thus, many individuals are availing themselves of the free testing services. LHWs will announce upcoming screening events in their community by advertising in Korean churches or Chinese language schools or by word-of-mouth. Our research team and LHWs will attend these events to recruit potential participants. Based on previous experiences, each screening event attracted about 100 to 150 Asian Americans. Second, the investigators will go to AAHC volunteer clinics to recruit participants every Saturday. About 10 to 12 Chinese or Korean patients visit the clinic. Patients usually come with family members. So, the investigators estimate to recruit about 15 to 20 participants at the clinics every Saturday. Finally, the investigators will identify potential participants by advertising in ethnic media and ethnic groceries.

Sample size estimate: Based on our previous studies (Juon et al. 2008; Hsu et al. 2007), the investigators estimate that about 10% of all the participants will test hepatitis B virus (HBV) positive, 40 to 50% will be HBV negative but protected, and about 50% will be unprotected. In the preliminary analysis of R25, there were significant mean differences of knowledge of HBV transmission (score ranged 0-10) in intervention (7.21±1.83SD) and control group (5.54±2.07SD) in post-test. The investigators estimated our sample size to be 50 in each intervention and control group among those unprotected. Assuming a conservative rate of attrition about 20%, the investigators calculated the study power based on sample size at follow-up. The sample size of 50 at pre-test is to detect mean difference in knowledge outcome at 96% power (1-β) and type I error of 0.05.Thus, our proposed sample size (n=50) for each group among those unprotected has sufficient power. Our total sample size is 600 (50/group x 2 groups x 2 (infected and protected-50% of study population) x 3 ethnic groups).

Specific Aim 3. To implement LHW intervention among those unprotected Procedures

1. Pre-test/Education program: After obtaining the informed consent for pre-test, screening test, and blood banking, all the participants will be asked to complete a self-administered questionnaire in English, Chinese, Korean, or Vietnamese, with the assistance of a bilingual interviewer when necessary. Then, LHW will provide a liver cancer education session to all participants in a small group setting.
2. HBV screening test/initial biospecimen banking: All participants will receive hepatitis B testing. For blood sampling procedure, the investigators will have a part-time phlebotomist working in the field with a bilingual staff and LHW. The phlebotomist will draw two tubes of blood from study participants at the study site. He/she will then transport one tube of the blood in red-top tube to certified clinical labs (i.e., Johns Hopkins Medical Institute (JHMI), Quest, LabCorp) for hepatitis B tests (e.g., HBsAg, HBsAb (surface antibody of HBV), HBcAb (core antibody of HBV)). The other tube will be processed for research sample banking.
3. Informing the results of screening test: All the participants will receive the results one week after their screening. Based on the screening results, all participants will be categorized into three groups: (1) infected (HbsAg+), (2) unprotected (HbsAg-/HbsAb-), and (3) protected (HbsAg-/HbsAb+). The investigators will order all screening tests and review all test results from the certified clinical labs. The investigators will mail the results to participants who are unprotected and protected. The investigators will not follow up healthy participants who are protected. The investigators will be responsible for informing the results by calling those infected individuals. The participants will provide counseling on what the results mean and treatment options.
4. Follow up for those infected: Those infected can either be referred through their primary care physicians to a hepatologist or directly to a hepatologist. If participants do not have a hepatologist, participants will be referred to hepatologists in the study team. This will be based on their language preference and geographic location.
5. LHW Intervention/follow up for those unprotected: Those unprotected will be randomly assigned to either the intervention or the control groups by computer-automated random assignment. Randomization will be used to assure equivalence between groups on key factors that may potentially influence the primary outcome of HBV vaccinations (e.g., gender, age, education, length of stay in the U.S.).

LHWs will conduct telephone interventions by reminding participants of a series of vaccinations at Months 1, 2, and 6 among those assigned to the intervention group. Those who have health insurance will be encouraged to complete vaccinations through their providers. If participants do not have health insurance, LHWs will provide resources to help those in the intervention access vaccinations by referring them to the AAHC, or County Health Departments who provide vaccinations to at risk populations. Those in the control group will receive a list of resources by mail that offers free vaccinations, such as local health departments along with their results. Upon completing follow-up, the investigators will provide the delayed LHW intervention for those who do not have vaccinations in the control group.

Seven months after mailing the results, those unprotected will be followed by phone to ask about their status of the series of vaccinations and promoters or barriers to vaccinations. Their self-reported vaccination will be verified with medical records. Participants will be asked to provide information about the date of vaccinations, as well as the location of the clinic or doctor's office where participants received vaccinations. Participants will also be asked to sign a medical release form giving project staff permission to request medical records for their vaccinations. The bilingual interviewers are blinded about participants being in the intervention or control group at post-test.

ELIGIBILITY:
Inclusion Criteria:

* foreign-born Asian American adults
* 18 years of age and older
* unprotected (HbsAg-/HbsAb-)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
self-reported status of the series of HBV vaccinations by follow-up calls in seven months after mailing the results verified by the medical records | Seven months after mailing the results
  Seven months after mailing the results, those unprotected were followed up by phone to ask about their status of the series of vaccinations and about promoters or barriers to vaccinations. Their self-reported vaccinations were verified with the medical records. Participants were asked to provide information about the date of vaccinations as well as the location of the clinic or doctor's office where participants received vaccinations. Participants were also asked to sign a medical release form giving project staff permission to request medical records regarding their vaccinations. Each participant was given a stamped vaccination card to fill out the date and provide the signature of their physician following each completed hepatitis B vaccination. Participants were asked to mail the card back to the research team once the card was completed.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soon Juon, PhD, Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson GF, Hussey PS. Population aging: a comparison among industrialized countries. Health Aff (Millwood). 2000 May-Jun;19(3):191-203. doi: 10.1377/hlthaff.19.3.191. PMID 10812799
- [Background] Caulfield LE, Gross SM, Bentley ME, Bronner Y, Kessler L, Jensen J, Weathers B, Paige DM. WIC-based interventions to promote breastfeeding among African-American Women in Baltimore: effects on breastfeeding initiation and continuation. J Hum Lact. 1998 Mar;14(1):15-22. doi: 10.1177/089033449801400110. PMID 9543954
- [Background] Earp JA, Viadro CI, Vincus AA, Altpeter M, Flax V, Mayne L, Eng E. Lay health advisors: a strategy for getting the word out about breast cancer. Health Educ Behav. 1997 Aug;24(4):432-51. doi: 10.1177/109019819702400404. PMID 9247823
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Han HR, Lee H, Kim MT, Kim KB. Tailored lay health worker intervention improves breast cancer screening outcomes in non-adherent Korean-American women. Health Educ Res. 2009 Apr;24(2):318-29. doi: 10.1093/her/cyn021. Epub 2008 May 7. PMID 18463411
- [Background] Hsu CE, Liu LC, Juon HS, Chiu YW, Bawa J, Tillman U, Li M, Miller J, Wang M. Reducing liver cancer disparities: a community-based hepatitis-B prevention program for Asian-American communities. J Natl Med Assoc. 2007 Aug;99(8):900-7. PMID 17722668
- [Background] Juon HS, Strong C, Oh TH, Castillo T, Tsai G, Oh LD. Public health model for prevention of liver cancer among Asian Americans. J Community Health. 2008 Aug;33(4):199-205. doi: 10.1007/s10900-008-9091-y. PMID 18363085
- [Background] Lefebvre RC, Flora JA. Social marketing and public health intervention. Health Educ Q. 1988 Fall;15(3):299-315. doi: 10.1177/109019818801500305. PMID 3056876
- [Background] Saunders RP, Evans MH, Joshi P. Developing a process-evaluation plan for assessing health promotion program implementation: a how-to guide. Health Promot Pract. 2005 Apr;6(2):134-47. doi: 10.1177/1524839904273387. PMID 15855283
- [Derived] Juon HS, Strong C, Kim F, Park E, Lee S. Lay Health Worker Intervention Improved Compliance with Hepatitis B Vaccination in Asian Americans: Randomized Controlled Trial. PLoS One. 2016 Sep 12;11(9):e0162683. doi: 10.1371/journal.pone.0162683. eCollection 2016. PMID 27617742